CLINICAL TRIAL: NCT01518660
Title: Multiple Sclerosis - Inflammatory, Neurological and Muscular Adaptations to Progressive Resistance Training
Brief Title: Multiple Sclerosis and Progressive Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS&PRT_SSAU_TK
Record Dates: First submitted 2012-01-06; First posted 2012-01-26 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2013-04

CONDITIONS: Multiple Sclerosis (Relapsing Remitting)
Keywords: Resistance Training; Strength Training
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Training (Experimental)
  Interventions: Behavioral: Training
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Training — Bi-weekly progressive resistance training
  Arms: Training

SUMMARY:
The purpose of this study is to investigate underlying mechanisms possibly explaining the beneficial effects of progressive resistance training for people with multiple sclerosis.

DETAILED DESCRIPTION:
Exercise in general, and progressive resistance training (PRT) in particular, is regarded as an important tool in the rehabilitation of people with multiple sclerosis (MS).

Previous studies have reported positive effects of PRT on muscle strength, functional capacity, fatigue and quality of life. Also, a possible disease modifying effect has been proposed. However, the underlying physiological mechanisms that might explain these beneficial effects and the possible effects on disease progression are unresolved. Additionally, none of the previous studies has been concerned with the possible impact of MS progression type, gender and/or medication.

The purpose of this randomized, controlled, gender stratified trial is to investigate underlying mechanisms possibly explaining the beneficial effects of progressive resistance training for people with multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed relapsing-remitting MS according to the McDonald criteria
* Expanded Disability Status Scale (EDSS) between 2.0 and 5.5
* Be able to train twice a week at the University
* Use interferon based medication

Exclusion Criteria:

* Alcohol abuse, Alzheimer's and pacemaker (or other metallic implant)
* Comorbidities like cardiovascular-, respiratory-, orthopaedic or metabolic diseases
* Having had an attack in a period of 8 weeks prior to the start of the intervention period
* Having an attack during the intervention period
* Pregnancy
* Systematic resistance training in a period of 3 months prior to the start of the intervention period.
* Training adherence of less than 85%.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Blood-borne biomarkers | Change from baseline to 24 weeks
  Resting levels of bloodbourne biomarkers;
  * Cytokines
  * Neurotrophins

SECONDARY OUTCOMES:
Neuro-muscular function of knee extensors | Change from baseline to 24 weeks
  By use of an isokinetic dynamometer, EMG and stimulation equipment the following will be assessed for the knee extensors;
  * Maximal muscle strength
  * Surface EMG
  * Central activation ratio
Walking performance | Change from baseline to 24 weeks
  Walking performance will be assessed by the;
  * Two minute walk test
  * 25-foot walk test
  * Chair rise test
  * Stair climb test
Self-reported measures | Change from baseline to 24 weeks
  The self-reported measures contains questionnaires regarding;
  * Fatigue (Fatigue Severity Scale, Modifies Fatigue Impact Scale)
  * Health-Related Quality of Life (SF-36)
  * Depression (Major Depression Inventory)
  * Disease impact (MS Impact Scale 29)
  * Walking Performance (MS Walking Scale 12)
Brain volume | Change from baseline to 24 weeks
  MRI-scans of the head will provide the following measurements;
  * Brain volume (analysed with SIENA)
  * Plaque incidence
Body Composition | Change from baseline to 24 weeks
  Weight and Bodyfat-% will be assessed with a Bodycomposition weight (Tanita SC220)
Thigh muscle cross-sectional area | Change from baseline to 24 weeks
  MRI-scans of the thigh will provide cross-sectional area of
  * m. quadriceps
  * m. hamstring

CONTACTS AND LOCATIONS:
Overall Officials: Tue Kjølhede, M.Sc., Principal Investigator — Sport Science, Department of Public Health, Aarhus University; Ulrik Dalgas, Ph.D., Study Chair — Sport Science, Department of Public Health, Aarhus University; Kristian Vissing, Ph.D., Study Chair — Sport Science, Department of Public Health, Aarhus University; Thor Petersen, Dr.med, Study Chair — MS Clinic, Department of Neurology, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - MS Clinic, Department of Neurology, Aarhus University Hospital, Aarhus C
  - Sport Science, Aarhus University, Aarhus C